CLINICAL TRIAL: NCT00858221
Title: Association of Genetic Variants in Obesity Genes to Resistance to Weight Loss and Susceptibility to Metabolic Syndrome in Morbidly Obese Patients: A Single Center, Blinded, Retrospective Clinical Study
Brief Title: Association of Genes to Resistance to Weight Loss in Obese Patients
Status: Completed | Type: Observational
Sponsor: Interleukin Genetics, Inc. (Industry)
Responsible Party: Karen Shaver, Director of Clinical Operations, Interleukin Genetics, Inc.
Other Study IDs: ILI-08-107PLIN
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Obesity; Metabolic Syndrome; Dyslipidemia
Keywords: obesity; genes; polymorphisms; weight loss; haplotype; diplotype
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Dyslipidemias; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA to be analyzed by genotyping
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall goal of this study is to determine whether variations in the perilipin, and several other, genes would be a useful tool for physicians who are caring for morbidly obese patients to guide therapy.

The main hypotheses to be tested is that sequence variations (polymorphisms) in the perilipin gene and several other obesity-related genes are associated with resistance to weight loss for obese individuals on energy restricted diets, potentially playing a role in the development of obesity related complications.

DETAILED DESCRIPTION:
The PRIMARY goal of this study is to investigate the association of perilipin gene polymorphisms, with obese subjects who are "resistant" to weight loss in a defined program.

The SECONDARY goal of this study is to investigate if additional candidate obesity genes that have previously been associated with obesity or energy metabolism show association with resistance to weight loss in subjects on an energy restricted diet. Additionally, we would like to investigate if any metabolic syndrome parameters, such as dyslipidemia or abnormal fasting glucose are associated with perilipin or variations in other obesity-related genes.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* competent patients interested in Gastric Bypass Surgery
* patients who are eligible for Gastric Bypass Surgery based on NIH criteria:

  * Male or Female
  * 21 - 70 years old, inclusive
  * Body Mass Index (BMI) > 40 with 2 co-morbid conditions such as Sleep Apnea, Hypertension, or Type 2 Diabetes
  * BMI > 45 with no co-morbid conditions

Exclusion Criteria:

* Patients not interested in Gastric Bypass Surgery
* Patients who do not qualify for surgery based on medical contraindications
* Patients with severe psychological contraindications
* Patients not willing to be compliant with pre-post surgical recommendations
* Patients younger than 21 years of age
* Patients older than 70 years of age
* Patients who do not qualify for surgery based on insurance constraints i.e., insurance guidelines for bypass surgery
* Patients who are pregnant
* Hispanic, Black, Asian Races
* Abnormal thyroid function

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian adults between the age of 21 and 70 years, inclusive, who fit the criteria for patients undergoing bariatric surgery at the Geisinger Clinic.
Sampling Method: Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Significant association of perilipin gene polymorphisms with obese subjects who are resistant to weight loss in a defined program. | 6 months

SECONDARY OUTCOMES:
Significant association of other genes, known to be obesity-related, with resistance to weight loss. Also, association of primary and secondary gene SNPs with dyslipidemia. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Shaver, MS, Study Director — Interleukin Genetics; Christopher D. Still, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States